CLINICAL TRIAL: NCT01711164
Title: The Role of FGL2-FcgammaRIIB Inhibitory Pathway in Human Viral Hepatitis
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-5129-BE
Record Dates: First submitted 2012-10-12; First posted 2012-10-22 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Hepatitis C Infection
Keywords: HCV; T regulatory cells (Tregs); FGL2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients: Chronic HCV patients who undergo antiviral therapy
- Healthy controls: healthy controls who are willing to give blood and liver tissue samples

SUMMARY:
Viral hepatitis is a serious world health problem affecting over 1 billion people worldwide. Presently the lack of highly effective treatments results in many patients requiring liver transplantation or death. The investigators have defined the role of a unique molecule FGL2 and its receptor fc-gammaR and its role in the pathogenesis of both experimental and human hepatitis. The studies proposed in the present proposal will test the hypothesis that measuring levels of fgl2 in plasma will identify individuals that will go on to develop chronic disease and inhibition of binding of fgl2 to its receptor will allow the host with both acute and chronic disease to develop an appropriate immune response and clear the virus. The studies will provide rationale for generation of new therapies to improve the treatment of patients with acute and chronic viral hepatitis by targeting fgl2.

DETAILED DESCRIPTION:
Hepatitis C Virus (HCV) infection affects more than 200 million individuals worldwide. Only a fraction of infected individuals clear the virus, whereas the majority (70%) develops chronic infection. The current standard of care, pegylated interferon/ ribavirin (pegIFN/rib) is effective in only 50% of patients. Patients who fail anti-viral therapy gradually progress to end-stage liver disease and hepatocellular cancer; which can only be cured by a liver transplant. The reasons for treatment failure are unclear but involve both viral and host factors. One significant factor may be impaired T cell function. Chronic HCV infection is associated with functionally impaired or exhausted cytotoxic T lymphocytes (CTLs), with decreased anti-viral cytokine production, cytotoxicity and proliferative capacity. The investigators recently showed that many patients who fail treatment have elevated frequencies of CD4+CD25+Foxp3+regulatory T cells (Tregs) producing the novel fibrinogen-like-protein 2 (FGL2/fibroleukin) which appears to impair HCV specific immune responses. Binding of FGL2 to the FcγRIIB receptor leads to inhibition of dendritic cell (DC) maturation, B cell apoptosis and inhibition of development of effective CD4+and CD8+T and B cell anti-viral responses. In HCV, increased levels of secreted FGL2 may suppress anti-viral immune responses and promote disease progression.

Hypothesis: HCV suppresses innate and adaptive anti-viral immune responses through the FGL2-FcγRIIB inhibitory pathway. Inhibition of this pathway will restore effective virus-specific immunity and lead to successful viral eradication.

Significance: These studies will establish the importance of FGL2-FcγRIIB inhibitory pathway in the pathogenesis of HCV chronic infection and provide a novel therapeutic approach to improve virus eradication and long term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Willing to follow the study protocol
3. Between >18 and <70 years of age, both gender
4. No history of active alcohol or drug abuse
5. Adequate contraception for both gender
6. Diagnosis of chronic HCV infection based on two positive serology tests.
7. Pre- and post treatment viral load data must be available
8. Naïve to antiviral treatment
9. A pre treatment liver biopsy should be available for all patients

Exclusion Criteria:

1. All other genotypes than genotype 1
2. Less than 18 or greater than 70 years of age
3. Pregnancy
4. Co-infection with HBV (hepatitis B virus), HDV (Hepatitis Delta virus) or HIV co-infection
5. Coexistence of liver disease of other etiology (autoimmune, alcohol)
6. Evidence of hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients being followed by hepatologists and considering treatment of Hepatitis C vs controls derived from potential live liver donors (for transplant)
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To correlate plasma levels of FGL2 in patients who undergo antiviral therapy for chronic HCV infection with clinical outcome | 6 months after end of antiviral treatment

SECONDARY OUTCOMES:
to correlate levels of FGL2 to numbers and immune function of CD4+ and CD8+ T cells, and DC activity | at all timepoints; pre-treatment, at wks 4, 12 and 48 of treatment and 6 months after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Selzner, MD PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Result] Foerster K, Helmy A, Zhu Y, Khattar R, Adeyi OA, Wong KM, Shalev I, Clark DA, Wong PY, Heathcote EJ, Phillips MJ, Grant DR, Renner EL, Levy GA, Selzner N. The novel immunoregulatory molecule FGL2: a potential biomarker for severity of chronic hepatitis C virus infection. J Hepatol. 2010 Oct;53(4):608-15. doi: 10.1016/j.jhep.2010.04.020. Epub 2010 Jun 17. PMID 20615566